CLINICAL TRIAL: NCT01484353
Title: Intensive Lifestyle Intervention for Type 2 Diabetics: The Kaiser Permanente TLC Pilot
Brief Title: Intensive Lifestyle Intervention for Type 2 Diabetics: The KP TLC Pilot
Acronym: KPTLCP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was cancelled.
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KPTLC Pilot
Record Dates: First submitted 2011-11-30; First posted 2011-12-02 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention group (Experimental): This is the only arm in the study. They will be compared before and after
  Interventions: Behavioral: Coronary Health Improvement Project Program

INTERVENTIONS:
Behavioral: Coronary Health Improvement Project Program — The Coronary Health Improvement Project' (CHIP; an intensive, community-based, lifestyle change program including a low saturated fat diet rich in whole, grown foods) has been shown to improve the health of diabetics through an intensive education taught over a 12 week period, but has not been studied in terms of its effect on HBAIC. Kaiser Permanente places significant resources into preventive medicine but does not have programs with the level of intensity of CHIP. This study aims to determine if Kaiser members with uncontrolled type 2 diabetes can achieve a significant improvement in their HBAIC after 12 weeks of participation in the CHIP program.

SUMMARY:
The purpose of this study is to determine if a healthy lifestyle intervention can significantly improve blood sugar control in type 2 diabetics over a course of 3 months.

DETAILED DESCRIPTION:
Peer reviewed research studies have proven the benefits of lifestyle interventions including the reversal of coronary artery disease and of diabetes. Experts agree that such a lifestyle must include a diet rich in whole, grown foods while low in saturated fat and cholesterol; regular physical activity; and healthy ways to cope with stress.

There are several challenges with implementing such lifestyle interventions such as educating the general public and health care providers to the components of this lifestyle and in getting people to adopt these healthy lifestyle changes.

While retreat-style, intensive lifestyle programs have shown that these obstacles can be overcome, they require monetary and time investments generally not feasible for the general public.

A community-based, lifestyle program such as 'The Coronary Health Improvement Project' program offers similar potential benefits at a more reasonable cost. It does so through an intensive education (32 hours total) taught over 4 weeks, followed by an 8-week consolidation period which include live or DVD based group sessions, discussions led by a program facilitator, and medical monitoring.

Kaiser Permanente, the leading Health maintenance organization in the nation, places special focus and significant resources into preventive medicine and health promotion, providing services to thousands of plan members but none with the level of intensity of 'The Coronary Health Improvement Project'.

This study aims to determine if 'The Coronary Health Improvement Project' program can significantly improve blood sugar control in kaiser plan members with uncontrolled diabetes.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking patients > 18 years of age, with at least 6 months of membership, who have type 2 diabetes.
* Patients must have a recent HbA1C lab value > 8.0, and have had at least 2 previous HbA1C measures during the previous 6-12 months.
* Patients with HbA1C values that are consistently > 8.0 over the previous 6-12 months will be invited to participate.

Exclusion Criteria:

1. current excessive alcohol use (drinking > 14 alcohol beverages per week for men or > 7 per week for women or > 4 per day for men or > 2 per day for women on 2 or more occasions each month)
2. current use of illegal or street drugs,
3. severely decreased functional capacity (shortness of breath or chest pain at rest or with minimal activity), and/or
4. suicidal thoughts or depression, will
5. Patients with severely limited physical ability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
HBAIC before and after intervention | 3 months
  Baseline HbA1C will be measured within two weeks of the start of the intervention. Follow-up HbA1C will be measured at 12 weeks after the start of the intervention, as HbA1C is a measure of glycemic control over approximately 12 weeks.

SECONDARY OUTCOMES:
Average weekly blood sugar | 3 months
  Baseline blood glucose readings will be checked one week prior to the start of the intervention, as well as weekly during the study for medication adjustment by a specialized Kaiser Permanente physician (weekly monitoring of blood glucose levels based on checks performed 3 times/day, for at least 3 consecutive days during the week, and then averaged). Follow-up blood glucose levels will be self-measured by patient glucometer, 3 times/ day, for at least 3 consecutive days. The average of these readings will be computed, as the "average weekly blood sugar"
Lipids | 3 months
  Baseline fasting lipid panel will be ascertained within two weeks prior to the start of the intervention. Follow-up fasting lipids will be measured at 4 weeks and at 12 weeks after the start of the intervention.
Weight | 3 months
  Baseline height, weight, waist circumference, hip circumference, and systolic and diastolic blood pressure will be measured within one week of the start of the intervention. Follow-up measures will be ascertained at 4, 8, and 12 weeks after the start of the intervention.
waist circumference | 3 months
  Baseline height, weight, waist circumference, hip circumference, and systolic and diastolic blood pressure will be measured within one week of the start of the intervention. Follow-up measures will be ascertained at 4, 8, and 12 weeks after the start of the intervention.
Blood pressure | 3 months
  Baseline height, weight, waist circumference, hip circumference, and systolic and diastolic blood pressure will be measured within one week of the start of the intervention. Follow-up measures will be ascertained at 4, 8, and 12 weeks after the start of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Mario A Robinson, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Riverside Medical Center, Riverside, California, United States